CLINICAL TRIAL: NCT04610931
Title: Study of the Effectiveness of a Virtual Reality Treatment in the Management of Smoking Cessation
Acronym: 3DSmoke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: National Cancer Institute, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RBHP 2020 BROUSSE
Record Dates: First submitted 2020-10-16; First posted 2020-11-02 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Tobacco Use Cessation
Keywords: Addiction; Tobacco; Virtual Reality Exposure Therapy; Cognitive Behaviour Therapy
MeSH Terms: conditions — Tobacco Use Cessation; Behavior, Addictive | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Random-sized block randomization, stratified on the number of previous relapses, will be performed for the inclusions of patients within the "cybertherapy" group or "Treatment as usual" group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cybertherapy (Experimental): use of cybertherapy (6 sessions) in addition to cognitive behavioral therapy (6 sessions) + pharmacological treatment
  Interventions: Behavioral: Virtual Reality-Enhanced Cognitive Behavioral Therapy (VR-CBT)
- Treatment as usual (Active Comparator): Treatment as usual is a cognitive behavioral therapy (6 sessions) + pharmacological treatment
  Interventions: Behavioral: cognitive behavior therapy

INTERVENTIONS:
Behavioral: Virtual Reality-Enhanced Cognitive Behavioral Therapy (VR-CBT) — Participants are smokers seeking treatment. Patients will be randomized into one of the 2 intervention groups.
  In all cases, patients will receive nicotine replacement therapy. The second physician in charge of the usual tobacco monitoring will adjust the dosage.
  Subjects in the usual treatment group will receive 6 weekly individual cognitive behavior therapy sessions lead by a psychologist. The content of CBT is similar in both groups. Subjects in the Virtual Reality group will receive 6 weekly individual CBT sessions followed by 6 virtual therapy sessions. Virtual therapy consists of exposing the patient to 3D situations considered to cause a high risk of smoking relapse and aiming to reduce signal reactivity by extinction. At each session, a neutral exposure will be given at the beginning to facilitate immersion and emergence of the session with a duration determined according to the sensitivity of each patient. Exposure is stopped when the craving approaches the baseline level.
  Arms: Cybertherapy
Behavioral: cognitive behavior therapy — Participants are smokers seeking treatment. Patients will be randomized into one of the 2 intervention groups. In all cases, patients will receive nicotine replacement therapy. The second physician in charge of the usual tobacco monitoring will adjust the dosage.
  Subjects in the usual treatment group will receive 6 weekly individual cognitive behavior therapy sessions lead by a psychologist. The content of CBT is similar in both groups.
  Arms: Treatment as usual

SUMMARY:
Tobacco is an addiction with serious consequences: somatic, psychiatric... The number of requests for treatment for tobacco addiction is gradually increasing from year to year, but conventional treatments have limited effectiveness. New tools such as virtual reality could be used in this treatment. We propose to create a virtual reality program based on the analysis of high-risk relapse situations. The investigator will then evaluate the effect of this cybertherapy on patients' relapse time and their desire to smoke.

DETAILED DESCRIPTION:
Smoking is the leading cause of morbidity and mortality, making it one of the most serious public health problems in the world. The majority of smokers would like to stop smoking and the number of smokers seeking treatment has increased by 25% between 2017 and 2018 in France. Indeed, many effective interventions have been developed to stop smoking, but many patients continue to relapse after a quit attempt. Only 10% to 30% achieve long-term abstinence and the majority relapse.

The therapeutic approach to addiction is based on a bio-psycho-social model. It aims to limit the runaway of subcortical processes (the cause of craving) via a medicinal approach and to strengthen the cortical control mechanisms via a psychotherapeutic approach.

As far as psychotherapeutic approaches are concerned, they seek to obtain a modification of cognitions and emotions related to tobacco through, for example, a relearning of the management of the product mediated by evocation or exposure. This may involve, for example, the repeated presentation (or evocation) of a signal (e.g. a place of consumption...), previously linked to consumption but in the absence of a reinforcer (product consumption). Most addiction remediation therapies have been developed and practiced with "imagination" (the patient is asked to think of stimulating situations) but they are difficult to control (because the patient's imagination can be more or less large) and are rarely used with situations that induce consumption. In this context the use of a 3Dimension (3D) tool, which allows a controlled and progressive exposure without confrontation, seems an interesting perspective. Virtual reality is recognized as a "tool" in the fields of neuroscience and psychology. It allows a patient-controlled exposure to complex, dynamic and three-dimensional stimuli.

Thus, virtual reality has logically been proposed as a tool in exposure therapies and its benefit has been measured in substance dependencies (Hone-Blanchet et al 2014). Since 2000, several researchers have successfully used virtual reality applications in addictions, but there is little data on objective evaluations of the effectiveness of cybertherapy in the treatment of tobacco addiction, particularly in association with the two reference treatments for smoking cessation that are nicotine substitution associated with cognitive behavioural therapy. For tobacco, the results are heterogeneous and did not take into account the different factors for maintaining tobacco use (Lee et al 2004, Choi et al 2011, Park et al 2014). Virtual therapy appears to be more effective when combined with other relapse prevention techniques such as cognitive behavioural therapy (CBT).

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 18 and 75 years of age
* Who smokes 10 or more cigarettes per day in the month prior to inclusion
* Who wants to quit smoking
* Who has a diagnosis of a smoking disorder with "craving" criteria according to DSM 5 criteria
* Who is able to speak and read French
* Who is covered by the French national health insurance system
* Who has a signed consent form

Exclusion Criteria:

* Subjects with decompensated psychiatric co-morbidities (DSM 5) or unstable organic disease
* Subjects at serious suicide risk
* Subjects with other substance use disorders (DSM 5)
* Problems that interact with 3D exposure: tendency to dissociation; interceptive phobias (panic attacks and hypochondria...); severe dizziness.
* Cognitive problems that limit or prevent the ability to implement coping strategies or the management of emotions or stimuli and disabilities to complete the questionnaires
* Subjects belonging to a protected population such as pregnant women, breastfeeding women, guardians
* Subjects deprived of liberty by judicial or administrative decision, subject to psychiatric treatment under duress, minor subject, or unable to express their consent
* Who refuses to participate

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2021-09-02 (Actual); Primary Completion 2026-01-07 (Actual); Study Completion 2026-01-07 (Actual)

PRIMARY OUTCOMES:
Percentage of patients who quit smoking | Day 43
  Comparison of proportion of patients who quit smoking after 6 weeks after intervention in the 2 arms (declarative status verified by measurement of carbon monoxide level in the expired air) and until one year.
Percentage of patients who quit smoking | Day 136
  Comparison of proportion of patients who quit smoking after 6 weeks after intervention in the 2 arms (declarative status verified by measurement of carbon monoxide level in the expired air) and until one year.
Percentage of patients who quit smoking | Day 229
  Comparison of proportion of patients who quit smoking after 6 weeks after intervention in the 2 arms (declarative status verified by measurement of carbon monoxide level in the expired air) and until one year.
Percentage of patients who quit smoking | Day 408
  Comparison of proportion of patients who quit smoking after 6 weeks after intervention in the 2 arms (declarative status verified by measurement of carbon monoxide level in the expired air) and until one year.

SECONDARY OUTCOMES:
smoking decreasing | Day 229, Day 408
  Comparison between arms of mean/median number of cigarette smoke per day (declarative status and measurement of carbon monoxide level in the expired air)
Craving score | Day 1, Day 43, Day 74, Day 136, Day 229, Day 408
  evaluation of craving score with Tabacco Craving Questionnary sort Form questionnaire (7 to 84; 7 no craving and 84 highest craving) ; comparison between arms at different endpoints
Needing score | Day 1, Day 43, Day 74, Day 136, Day 229, Day 408
  It is evaluated with an analogical visual scale (1 to 10; 1 the lowest 10 the highest); comparison between arms at different endpoints
e-health score | Day 1, Day 43
  It is evaluated with disease simulation questionnaire (French Speach Spatial en Quality -SSQ-vf- questionnaire)(/16)
Follow-up of all virtual reality sessions | Day 43
  Follow-up of all virtual reality sessions is assessed at 6 weeks post-inclusion
Relapse rate | Day 1, Day 43, Day 74, Day 136, Day 229, Day 408
  Relapse rate is the percentage of participants who are abstinent at the end of treatment and who relapse during the follow-up period; comparison between arms at different endpoints
Level of anxiety and depression | Day 1, Day 43, Day 74, Day 136, Day 229, Day 408
  It is evaluated with the Hospital Anxiety and Depression - HAD scale (1 to 21; 1 no anxiety and depression , 21 highest symptoms); comparison between arms at different endpoints

CONTACTS AND LOCATIONS:
Locations (1):
- Clermont-Ferrand University Hospital, Clermont-Ferrand, Auvergne, France